CLINICAL TRIAL: NCT04223050
Title: Will Titrated Oxygen Flow to a Peripheral Oxygen Saturation of 88-92% Compared With Oxygen Flow to a Saturation >94% Reduce Mortality in Chronic Obstructive Pulmonary Disease Patients With Acute Exacerbation? - a Randomized Clinical Trial
Brief Title: Comparing Mortality for Low vs High Peripheral Oxygen Saturation in COPD-patients With Acute Exacerbation
Acronym: O2flow-COPD
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Esbjerg Hospital - University Hospital of Southern Denmark (Other)
Collaborators: Holbaek Sygehus (Other); Odense University Hospital (Other); Sygehus Lillebaelt (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2019-002498-80; 19/4298 (Registry Identifier: Region of Southern Denmark); 2019-002498-80 (EudraCT Number)
Record Dates: First submitted 2020-01-07; First posted 2020-01-10 (Actual); Last update posted 2022-11-01 (Actual); Status verified 2022-10

CONDITIONS: COPD Exacerbation; Chronic Obstructive Pulmonary Disease Exacerbation
Keywords: COPD; Oxygen treatment; Mortality
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — nitrox

STUDY DESIGN:
Intervention Model Description: Randomization will be performed as block randomization with a 1:1 allocation using an electronic randomization system accessible via the internet (REDCap via OPEN at the University of Southern Denmark). The participants will be randomized electronically bedside by the study representatives.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- High oxygen saturation (Active Comparator): Peripheral oxygen saturation level >94%
  Interventions: Drug: Oxygen gas
- Low oxygen saturation (Active Comparator): Peripheral oxygen saturation level 88-92%
  Interventions: Drug: Oxygen gas

INTERVENTIONS:
Drug: Oxygen gas — Administering oxygen to achieve the desired peripheral oxygen saturation

SUMMARY:
Chronic obstructive pulmonary disease (COPD) is a common disorder that affects approximately 400,000 Danish citizens. About 3,000-3,500 Danes die yearly because of the disorder, and the costs associated with hospital admissions are estimated to be 535 million Danish kroner (DKK). Patients with COPD risk a worsening of their disorder, and in most cases, this will require hospitalization. One of the used treatments is providing oxygen to the patients via e.g. masks. The recommendations on oxygen treatment are currently based on a study from 2010 where 37% of the participants in this study did not receive the intended treatment, which may have had massive effects on the results. It is worrying that no other studies have shown which oxygen treatment is safest for the patients. As such, we deem it important to study how best to treat the patients.

Our study is of high clinical relevance as hospitals receive patients with worsening of COPD daily. We need more, better data regarding the oxygen treatment of our patients, in order to provide our patients with the best possible care. The purpose of our study is thus to determine which oxygen treatment is best for patients with acute worsening of COPD symptoms. We will use a prospective, randomized controlled open-label trial. We will use two treatments: Treatment 1 is giving oxygen to the patient to reach a peripheral oxygen saturation of above 94%. Treatment 2 is giving oxygen to reach a peripheral oxygen saturation of between 88% and 92%.

Our primary outcome is 30-day all-cause mortality, with secondary outcomes being 7-day all-cause mortality, need for non-invasive ventilation, intubation or intensive care admission, over-all length of hospital stay and respiratory acidosis.

We believe that a lower oxygen saturation percentage may be superior as one study (Austin et al., 2010) showed a lower mortality rate in the group of patients that had a lower peripheral oxygen saturation. Additionally, the risk of respiratory acidosis and hypercapnia were lower. We wish to perform our study in the hospital sector as this study was performed in the prehospital sector and thus their results cannot be translated directly.

DETAILED DESCRIPTION:
Please refer to the full protocol.

ELIGIBILITY:
Inclusion Criteria:

* age 18 years or older
* ability to give informed consent
* previously diagnosed COPD (either confirmed diagnosis at prior hospital - contact or from their general practitioner or confirmed diagnosis by the treating physician in the emergency department (verified by use of relevant medication))
* admitted with acute exacerbation (acute and worsened shortness of breath) of COPD
* requiring oxygen treatment

Exclusion Criteria:

* Instability at arrival requiring immediate lifesaving treatment, e.g. intubation or non-invasive ventilation, within the first 30 minutes
* Expected total length of stay in hospital < 12 hours
* Planned transfer to another hospital within 12 hours
* Unwilling to have repeated arterial blood gas analyses within the first 12 hours
* Patients judged terminal by treating physician in the emergency department
* Non-residents of the particular country
* Expected impossible follow-up
* Fertile women (<50 years of age) with positive urine human gonadotropin (hCG) or plasma-hCG
* Prior participation in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 415 (Estimated)
Dates: Start 2020-02-03 (Actual); Primary Completion 2024-08-31 (Estimated); Study Completion 2024-08-31 (Estimated)

PRIMARY OUTCOMES:
30-day all-cause mortality | 30 days
  Data is extracted from the Danish national registries.

SECONDARY OUTCOMES:
7-day all-cause mortality | 7 days
  Data is extracted from the Danish national registries.
Non-invasive ventilation | 12 hours
  The Medical records will be reviewed for documentation on if the patient has been on non-invasive ventilation. This will be reported as proportion of patients on NIV
Intubation | 12 hours
  The Medical records will be reviewed for documentation on if the patient has been intubated. This will be reported as proportion of patients intubated
Intensive care admission | 1 day
  Extracted from the hospital records.
Overall length of hospital stay | 10 days
  Time calculated from the hospital records
Respiratory acidosis | 12 hours
  Measured as an arterial blood gas analysis with pH > 7.35 and hypercapnia

CONTACTS AND LOCATIONS:
Overall Officials: Peter Hallas, MD, Principal Investigator — Holbaek Sygehus; Sune Laugesen, MD, Principal Investigator — Odense University Hospital; Simon Thorgaard-Rasmussen, MD, Principal Investigator — Sygehus Lillebælt, Kolding
Locations (4):
- Denmark (4):
  - Sydvestjysk Sygehus, Esbjerg
  - Holbæk Sygehus, Holbæk
  - Sygehus Lillebælt, Kolding, Kolding
  - Odense University Hospital, Odense

IPD SHARING:
Plan to Share IPD: No
(Indsæt senere)